CLINICAL TRIAL: NCT01050036
Title: Phase 2 Study of Autologous Hematopoietic Cell Transplantation for Core-binding Factor Positive Acute Myeloid Leukemia in the First Complete Remission
Brief Title: Autologous Hematopoietic Cell Transplantation for Core-binding Factor Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Je-Hwan Lee, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-H-54
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Myeloid
Keywords: Leukemia, Myeloid; Primary complete remission; Favorable karyotype; Autologous hematopoietic cell transplantation; Hematopoietic cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCT recipients (Experimental): 1. Patient with CBF AML will be eligible in his/her 1st complete remission (CR1) status. Patients who have relapsed or have achieved 2nd complete remission should not be included in this study.
  2. 1st postremission therapy after CR1 will be performed with high-dose cytarabine (HDAC) chemotherapy, consisting of intravenous cytarabine 3 g/m2 infusion during 3 hours twice a day on days 1, 3, and 5.
  3. After achieving CR1, patient will be invited to this protocol and will be able to decide whether to join or not after listening to the information.
  Interventions: Procedure: autologous hematopoietic cell transplantation

INTERVENTIONS:
Procedure: autologous hematopoietic cell transplantation — 1. Autologous peripheral blood stem cell (PBSCs) harvesting
     * After the second cycle of high-dose ara-C(HDAC) consolidation chemotherapy
     * Mobilization: recombinant human G-CSF(Filgrastim) 5mcg/kg s.c. daily starting on 10 days after start of the second cycle of HDAC chemotherapy
     * Harvest procedure: peripheral blood mononuclear cells will be collected. Target CD34+ cell dose is over 5x10E6/kg.
  2. Conditioning regimen for autologous HCT
     * Busulfan 3.2 mg/kg/day i.v. daily on days -7 to -5 (for 3 days)
     * Etoposide 400mg/m2/day i.v. daily on days -3 to -2 (for 2 days)
  3. Autologous cell infusion and waiting for engraftment
  Other Names: Busulfex; Etoposid; Grasin

SUMMARY:
Primary study objective is the evaluation of efficacy of autologous hematopoietic cell transplantation (HCT) with core-binding factor (CBF) positive acute myeloid leukemia (AML) in the first CR (CR1) in terms of relapse incidence (cumulative incidence of relapse, CIR) and disease-free survival (DFS).

Secondary study objectives are the engraftment rate / time to engraftment, transplantation-related mortality (TRM) rate, event-free survival (EFS) rate, and Overall survival (OS).

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE 1.1. CLINICAL CHARACTERISTICS OF CBF AML Acute myeloid leukemia (AML) is a disease entity consisting of heterogeneous groups with different clinical features and prognosis. Cytogenetic status of patients with AML is the single most important factor to expect the survival and the treatment responses.

Core binding factor (CBF) AML is characterized by the presence of cytogenetic abnormalities, i.e., the balanced translocation between chromosome 8 and 21 [t(8;21)(q22;q22)] and the pericentric inversion of chromosome 16 [inv(16)(p13q22)] or its less frequent variant, the balanced translocation t(16;16)(p13;q22). Among adults with de novo AML, t(8;21) and inv(16) are found in 7% and 8% of patients, respectively1. All the subtypes of CBF AML share the same chimeric fusion genes that are formed by the disruption of genes encoding different subunits of the core binding factor, a heterodimeric transcription factor complex.

CBF AML has been accepted as a disease entity of favorable prognosis with a high complete remission rate (up to 90%) with conventional induction chemotherapy followed by an intensive consolidation treatment of 3 or 4 cycles of high-dose cytarabine(HDAC). The overall survival of patients in this group rise up to 60 - 70 %, and this encouraging result has supported the opinion that HDAC was a more preferable postremission therapy instead of autologous hematopoietic cell transplantation (HCT) or allogeneic HCT.

1.2. STRATEGY TO REDUCE RELAPSE IN CBF AML It has been thought that patients with CBF AML in first complete remission (CR1) would benefit most from high-dose consolidation chemotherapy and the risk of HCT outweigh the benefit in this group. However, the cumulative incidence of relapse (CIR) has been reported to be up to 54% and 50-60% of patients are cured using contemporary treatment. The survival outcome is unsatisfactory, especially in elderly patients. Prebet et al reported that the 5-year probabilities of overall survival (OS) and leukemia-free survival (LFS) were 31% and 27%, respectively with intensive consolidation or low-dose maintenance chemotherapy among patients with CBF AML who were age 60 years or older. To improve the treatment outcome in this group, alternative strategies of postremission therapy with more efficiency and more tolerability are warranted, especially for patients who are prone to relapse. A number of studies about the stratified intensification of postremission therapy according to the risk of relapse and the appropriate prognostic index for identifying high risk patients have been reported, and some of them are currently under investigation.

1.3. DIFFERENCES BETWEEN AML WITH INV(16) AND WITH T(8;21) Recent studies have reported that these two groups seem to be distinct clinical entities and should be stratified and reported separately. Patients with t(8;21) had shorter OS (hazard ratio [HR] =1.5, p=0.045) and survival after first relapse (HR=1.7, p=0.009) than patients with inv(16). A similar difference was found among patients who had undergone HCT; the 3-year OS of patients with t(8;21) and inv(16) was 50% and 72%, respectively(p=0.002). Based on these results, a discriminative postremission strategy could be applied to patients with CBF AML - patients with t(8;21) should be managed differently from those with inv(16) as to the application of HCT and a prospective trial can be warranted to clarify the significance of HCT over chemotherapy.

1.4. RISK STRATIFICATION IN AML WITH INV(16) Although AML with inv(16) has a relatively good prognosis, a substantial number of these patients (i.e. 40-50%) finally relapse. In this group, timely identification and therapeutic stratification of patients who deemed at high risk for relapse could ultimately result in an improvement of clinical outcomes. The minimal residual disease (MRD) monitoring with real-time quantitative polymerase chain reaction (RQ-PCR) assays for CBFβ/MYH11 fusion transcript has been regarded as a useful surrogate marker for identifying a patient with resistant disease and for predicting relapse early during remission. Lane et al reported that a rise of the same or more than 1 log rise of transcript level relative to the level from a remission bone marrow sample at any time of post-induction follow up correlated with inferior LFS and morphologic relapse (HR 8.6). Bounamici et al suggested that patients whose transcript ratios of bone marrow samples taken during remission were greater than 0.25% finally relapse, and ratio below 0.12% might indicate that patients is in a curable state.

Two conclusions can be deduced from the results above; first, a considerable portion of patients among those with CBF AML finally relapse. Second, post-induction MRD monitoring might be helpful in discriminating patients who are vulnerable to relapse and may have benefit with more intensified consolidation therapy.

1.5. RISK STRATIFICATION IN AML WITH T(8;21) AML with t(8;21) has been accepted as a disease of good prognosis and categorized to favorable cytogenetic risk group along with AML with inv(16). According to recent studies, however, outcomes of AML patients with t(8;21) were disappointing in contrary to those with previous ones. The biologic and prognostic heterogeneity have been recently described for this subgroup (including other subtypes of CBF AML) and a number of promising biologic markers have been suggested.

MRD monitoring with RQ-PCR or flow cytometry is also thought as a useful method for the stratification of patients with t(8;21), as well as for those with inv(16). C-kit mutation has been generally accepted as a discriminating marker of CBF AML which increase the relapse risk. A difference in race has been considered as an important predictor for t(8;21) AML, in that nonwhites failed induction more often and had shorter OS than white. Other biomarkers which has been being considered are leukocyte count or white blood cell, CD56 positivity, loss of sex chromosome and secondary cytogenetic abnormalities6, submicroscopic deletion during chromosome rearrangement, loss of MRP gene during translocation / inversion and presence of RAS/FLT3 mutation. Gene-expression profile is suggested as a relevant way of molecular characterization to discriminate substantial biologic and clinical heterogeneity within CBF AML.

1.6. COMPARISON OF POSTREMISSION THERAPY FOR CBF AML The optimal postremission therapy of CBF AML remains to be determined. Despite being considered as patients in more favorable risk group in AML, only approximately half of the patients are cured with current strategy, significant portion of patients finally relapse and the overall survival is unsatisfactory. Heterogeneity of the treatment outcome in this group also suggests that a tailored approach might be preferred to a unique predefined strategy to treat. Current state of CBF AML indicates the need for improved therapeutic approaches, including more intensive consolidation to obtain improved LFS.

There were a few prospective studies that support the role of HCT. A prospective trial on the impact of cytogenetics and the kind of consolidation therapy performed by Visani et al showed that patients in the favorable group had significantly longer disease-free survival(DFS) when treated with an intensive induction and allogeneic HCT as an intensive consolidation therapy. According to the result of MRC AML 10 randomized controlled trial comparing the addition of autologous HCT with intensive chemotherapy alone for AML in CR1, addition of autologous HCT to four course of intensive chemotherapy reduced the risk of relapse, increased disease-free survival significantly, and improved the overall survival, although there were more death in remission in the autologous HCT group. However, a number of studies support the classic concept that CBF AML in CR1 would benefit most from HDAC and the risk of HCT outweigh the benefit. Delaunay et al reported that outcome of patients with inv(16) in CR1 was similar among patients allocated to receive allogeneic HCT vs HDAC8. According to the meta-analysis performed on 392 adults with CBF AML in prospective German AML treatment trial, type of postremission therapy revealed no difference between intensive chemotherapy and autologous HCT in the t(8;21) group and between chemotherapy, autologous HCT, and allogeneic HCT in the inv(16) group. Recent results suggest the possibility of improving overall survival with HCT. Subgroup analysis of EORTC-LG/GIMEMA AML-10 trial in which patients younger than 46 years were assigned to allogeneic HCT or autologous HCT according to the availability of HLA-identical sibling donor, DFS rate were similar in patients with good risk cytogenetics. Kuwatsuka et al reported a retrospective analysis on the results of HCT performed on CBF AML. OS was not different between patients in CR1 who received allogeneic HCT and those who received autologous HCT for both t(8;21) AML (84% vs 77%; p=0.49) and inv(16) AML (74% vs 59%, p=0.86).

1.7. OPTIMAL POSTREMISSION THERAPY FOR CBF AML In summary, HDAC chemotherapy has been recommended as a relevant postremission therapy for patients with CBF AML in CR1 on the basis that risk of HCT outweigh the clinical benefit of reducing the incidence of relapse and prolonging LFS. With the advances in hematopoietic cell transplantation technique and biomarkers for risk stratification, HCT is now considered for a promising method to improve the overall outcome of patients with CBF AML. Until now, previous results support the introduction of autologous HCT rather than allogeneic HCT for intensified postremission therapy in CBF AML in that the benefit of HCT was not yet proven and the risk of allogeneic HCT might outweigh the benefit in this group. We hereby intend to evaluate the efficacy of autologous HCT in patients with CBF AML in CR1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CBF positive AML in CR1. CBF AML includes t(8;21)(q22;q22) [AML1(RUNX1)/ETO(CBFα2T1)], inv(16)(q13q22) (CBFβ/MYH11), t(16;16)(p13;q22) (CBFβ/MYH11) Using RT-PCR, FISH, or standard karyotype analysis technique.
* Patients who plan to receive the second cycle of HDAC consolidation chemotherapy.
* 15 years old or older and 65 years or younger
* Adequate performance status (Karnofsky score of 70 or more).
* Adequate hepatic and renal function (AST, ALT, and bilirubin < 3.0 x upper normal limit, and creatinine < 2.0 mg/dL).
* Adequate cardiac function (left ventricular ejection fraction over 40% on heart scan or echocardiography)
* Signed and dated informed consent must be obtained from patient.

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01-11 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of relapse | 3 years
  cumulative incidence of relapse

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  defined as the interval between the day when complete remission is confirmed with bone marrow biopsy report (not by the day when bone marrow biopsy was performed) and the day when the relapse is confirmed by bone marrow biopsy or the presence of peripheral blood.
engraftment rate | 100 days
  defined as the interval between day 0 (PBSCs infusion) and the first day of evidence for engraftment.
transplantation-related mortality | 100 days
  transplantation-related mortality
Event-free survival | 3 years
  defined as the interval between day 0-PBSCs infusion and the event.
Overall survival | 3 years
  measured from day 0 to the date of last follow-up or death.

CONTACTS AND LOCATIONS:
Overall Officials: Je-Hwan Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (11):
- South Korea (11):
  - Wonkwang University Hospital, Iksan, Chollabuk-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Hallym University Sacred Heart Hospital, Anyang, Kyeongki-do
  - Kosin University, Gospel Hospital, Busan
  - Busan Paik Hospital, Inje University College of Medicine, Busan
  - Daegu Fatima Hospital, Daegu
  - Yeongnam University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Gachon University Gil Hospital, Inchon
  - Asan Medical Center, Seoul
  - Ulsan University Hospital, University of Ulsan College of Medicine, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrd JC, Mrozek K, Dodge RK, Carroll AJ, Edwards CG, Arthur DC, Pettenati MJ, Patil SR, Rao KW, Watson MS, Koduru PR, Moore JO, Stone RM, Mayer RJ, Feldman EJ, Davey FR, Schiffer CA, Larson RA, Bloomfield CD; Cancer and Leukemia Group B (CALGB 8461). Pretreatment cytogenetic abnormalities are predictive of induction success, cumulative incidence of relapse, and overall survival in adult patients with de novo acute myeloid leukemia: results from Cancer and Leukemia Group B (CALGB 8461). Blood. 2002 Dec 15;100(13):4325-36. doi: 10.1182/blood-2002-03-0772. Epub 2002 Aug 1. PMID 12393746
- [Background] Burgess JK, Lopez JA, Berndt MC, Dawes I, Chesterman CN, Chong BH. Quinine-dependent antibodies bind a restricted set of epitopes on the glycoprotein Ib-IX complex: characterization of the epitopes. Blood. 1998 Oct 1;92(7):2366-73. PMID 9746776
- [Background] Slovak ML, Kopecky KJ, Wolman SR, Henslee-Downey JP, Appelbaum FR, Forman SJ, Blume KG. Cytogenetic correlation with disease status and treatment outcome in advanced stage leukemia post bone marrow transplantation: a Southwest Oncology Group study (SWOG-8612). Leuk Res. 1995 Jun;19(6):381-8. doi: 10.1016/0145-2126(94)00162-4. PMID 7596150
- [Background] Paschka P. Core binding factor acute myeloid leukemia. Semin Oncol. 2008 Aug;35(4):410-7. doi: 10.1053/j.seminoncol.2008.04.011. PMID 18692691
- [Background] Speck NA, Gilliland DG. Core-binding factors in haematopoiesis and leukaemia. Nat Rev Cancer. 2002 Jul;2(7):502-13. doi: 10.1038/nrc840. No abstract available. PMID 12094236
- [Background] Marcucci G, Mrozek K, Ruppert AS, Maharry K, Kolitz JE, Moore JO, Mayer RJ, Pettenati MJ, Powell BL, Edwards CG, Sterling LJ, Vardiman JW, Schiffer CA, Carroll AJ, Larson RA, Bloomfield CD. Prognostic factors and outcome of core binding factor acute myeloid leukemia patients with t(8;21) differ from those of patients with inv(16): a Cancer and Leukemia Group B study. J Clin Oncol. 2005 Aug 20;23(24):5705-17. doi: 10.1200/JCO.2005.15.610. PMID 16110030
- [Background] Schlenk RF, Benner A, Krauter J, Buchner T, Sauerland C, Ehninger G, Schaich M, Mohr B, Niederwieser D, Krahl R, Pasold R, Dohner K, Ganser A, Dohner H, Heil G. Individual patient data-based meta-analysis of patients aged 16 to 60 years with core binding factor acute myeloid leukemia: a survey of the German Acute Myeloid Leukemia Intergroup. J Clin Oncol. 2004 Sep 15;22(18):3741-50. doi: 10.1200/JCO.2004.03.012. Epub 2004 Aug 2. PMID 15289486
- [Background] Delaunay J, Vey N, Leblanc T, Fenaux P, Rigal-Huguet F, Witz F, Lamy T, Auvrignon A, Blaise D, Pigneux A, Mugneret F, Bastard C, Dastugue N, Van den Akker J, Fiere D, Reiffers J, Castaigne S, Leverger G, Harousseau JL, Dombret H; French Acute Myeloid Leukemia Intergroup; Groupe Ouest-Est des Leucemies Aigues Myeoblastiques; Leucemies Aigues Myeoblastiques de l'Enfant; Acute Leukemia French Association; Bordeaux-Grenoble-Marseille-Toulouse cooperative groups. Prognosis of inv(16)/t(16;16) acute myeloid leukemia (AML): a survey of 110 cases from the French AML Intergroup. Blood. 2003 Jul 15;102(2):462-9. doi: 10.1182/blood-2002-11-3527. Epub 2003 Mar 20. PMID 12649129
- [Background] Perea G, Lasa A, Aventin A, Domingo A, Villamor N, Queipo de Llano MP, Llorente A, Junca J, Palacios C, Fernandez C, Gallart M, Font L, Tormo M, Florensa L, Bargay J, Marti JM, Vivancos P, Torres P, Berlanga JJ, Badell I, Brunet S, Sierra J, Nomdedeu JF; Grupo Cooperativo para el Estudio y Tratamiento de las Leucemias Agudas y Miel. Prognostic value of minimal residual disease (MRD) in acute myeloid leukemia (AML) with favorable cytogenetics [t(8;21) and inv(16)]. Leukemia. 2006 Jan;20(1):87-94. doi: 10.1038/sj.leu.2404015. PMID 16281071
- [Background] Appelbaum FR, Kopecky KJ, Tallman MS, Slovak ML, Gundacker HM, Kim HT, Dewald GW, Kantarjian HM, Pierce SR, Estey EH. The clinical spectrum of adult acute myeloid leukaemia associated with core binding factor translocations. Br J Haematol. 2006 Oct;135(2):165-73. doi: 10.1111/j.1365-2141.2006.06276.x. Epub 2006 Aug 25. PMID 16939487
- [Background] Prebet T, Boissel N, Reutenauer S, Thomas X, Delaunay J, Cahn JY, Pigneux A, Quesnel B, Witz F, Thepot S, Ugo V, Terre C, Recher C, Tavernier E, Hunault M, Esterni B, Castaigne S, Guilhot F, Dombret H, Vey N; Acute Leukemia French Association; Groupe Ouest-Est des leucemies et autres maladies du sang (GOELAMS); Core Binding Factor Acute Myeloid Leukemia (CBF AML) intergroup. Acute myeloid leukemia with translocation (8;21) or inversion (16) in elderly patients treated with conventional chemotherapy: a collaborative study of the French CBF-AML intergroup. J Clin Oncol. 2009 Oct 1;27(28):4747-53. doi: 10.1200/JCO.2008.21.0674. Epub 2009 Aug 31. PMID 19720919
- [Background] Mrozek K, Marcucci G, Paschka P, Bloomfield CD. Advances in molecular genetics and treatment of core-binding factor acute myeloid leukemia. Curr Opin Oncol. 2008 Nov;20(6):711-8. doi: 10.1097/CCO.0b013e32831369df. PMID 18841055
- [Background] Kuwatsuka Y, Miyamura K, Suzuki R, Kasai M, Maruta A, Ogawa H, Tanosaki R, Takahashi S, Koda K, Yago K, Atsuta Y, Yoshida T, Sakamaki H, Kodera Y. Hematopoietic stem cell transplantation for core binding factor acute myeloid leukemia: t(8;21) and inv(16) represent different clinical outcomes. Blood. 2009 Feb 26;113(9):2096-103. doi: 10.1182/blood-2008-03-145862. Epub 2009 Jan 6. PMID 19126873
- [Background] Picard C, Silvy M, Gabert J. Overview of real-time RT-PCR strategies for quantification of gene rearrangements in the myeloid malignancies. Methods Mol Med. 2006;125:27-68. doi: 10.1385/1-59745-017-0:27. PMID 16502577
- [Background] Lane S, Saal R, Mollee P, Jones M, Grigg A, Taylor K, Seymour J, Kennedy G, Williams B, Grimmett K, Griffiths V, Gill D, Hourigan M, Marlton P. A >or=1 log rise in RQ-PCR transcript levels defines molecular relapse in core binding factor acute myeloid leukemia and predicts subsequent morphologic relapse. Leuk Lymphoma. 2008 Mar;49(3):517-23. doi: 10.1080/10428190701817266. PMID 18297529
- [Background] Buonamici S, Ottaviani E, Testoni N, Montefusco V, Visani G, Bonifazi F, Amabile M, Terragna C, Ruggeri D, Piccaluga PP, Isidori A, Malagola M, Baccarani M, Tura S, Martinelli G. Real-time quantitation of minimal residual disease in inv(16)-positive acute myeloid leukemia may indicate risk for clinical relapse and may identify patients in a curable state. Blood. 2002 Jan 15;99(2):443-9. doi: 10.1182/blood.v99.2.443. PMID 11781223
- [Background] Lee KW, Choi IS, Roh EY, Kim DY, Yun T, Lee DS, Yoon SS, Park S, Kim BK, Kim NK. Adult patients with t(8;21) acute myeloid leukemia had no superior treatment outcome to those without t(8;21): a single institution's experience. Ann Hematol. 2004 Apr;83(4):218-24. doi: 10.1007/s00277-003-0811-1. Epub 2003 Nov 20. PMID 14628154
- [Background] Ma SK, Au WY, Kwong YL, Lam CK, Liang RH, Chan LC. Hematological features and treatment outcome in acute myeloid leukemia with t(8;21). Hematol Oncol. 1997 May;15(2):93-103. doi: 10.1002/(sici)1099-1069(199705)15:23.0.co;2-g. PMID 9375034
- [Background] Leroy H, de Botton S, Grardel-Duflos N, Darre S, Leleu X, Roumier C, Morschhauser F, Lai JL, Bauters F, Fenaux P, Preudhomme C. Prognostic value of real-time quantitative PCR (RQ-PCR) in AML with t(8;21). Leukemia. 2005 Mar;19(3):367-72. doi: 10.1038/sj.leu.2403627. PMID 15674426
- [Background] Marcucci G, Caligiuri MA, Bloomfield CD. Core binding factor (CBF) acute myeloid leukemia: is molecular monitoring by RT-PCR useful clinically? Eur J Haematol. 2003 Sep;71(3):143-54. doi: 10.1034/j.1600-0609.2003.00131.x. PMID 12930314
- [Background] Yin JA, Frost L. Monitoring AML1-ETO and CBFbeta-MYH11 transcripts in acute myeloid leukemia. Curr Oncol Rep. 2003 Sep;5(5):399-404. doi: 10.1007/s11912-003-0026-6. PMID 12895392
- [Background] Paschka P, Marcucci G, Ruppert AS, Mrozek K, Chen H, Kittles RA, Vukosavljevic T, Perrotti D, Vardiman JW, Carroll AJ, Kolitz JE, Larson RA, Bloomfield CD; Cancer and Leukemia Group B. Adverse prognostic significance of KIT mutations in adult acute myeloid leukemia with inv(16) and t(8;21): a Cancer and Leukemia Group B Study. J Clin Oncol. 2006 Aug 20;24(24):3904-11. doi: 10.1200/JCO.2006.06.9500. PMID 16921041
- [Background] Boissel N, Leroy H, Brethon B, Philippe N, de Botton S, Auvrignon A, Raffoux E, Leblanc T, Thomas X, Hermine O, Quesnel B, Baruchel A, Leverger G, Dombret H, Preudhomme C; Acute Leukemia French Association (ALFA); Leucemies Aigues Myeloblastiques de l'Enfant (LAME) Cooperative Groups. Incidence and prognostic impact of c-Kit, FLT3, and Ras gene mutations in core binding factor acute myeloid leukemia (CBF-AML). Leukemia. 2006 Jun;20(6):965-70. doi: 10.1038/sj.leu.2404188. PMID 16598313
- [Background] Care RS, Valk PJ, Goodeve AC, Abu-Duhier FM, Geertsma-Kleinekoort WM, Wilson GA, Gari MA, Peake IR, Lowenberg B, Reilly JT. Incidence and prognosis of c-KIT and FLT3 mutations in core binding factor (CBF) acute myeloid leukaemias. Br J Haematol. 2003 Jun;121(5):775-7. doi: 10.1046/j.1365-2141.2003.04362.x. PMID 12780793
- [Background] Nguyen S, Leblanc T, Fenaux P, Witz F, Blaise D, Pigneux A, Thomas X, Rigal-Huguet F, Lioure B, Auvrignon A, Fiere D, Reiffers J, Castaigne S, Leverger G, Harousseau JL, Socie G, Dombret H. A white blood cell index as the main prognostic factor in t(8;21) acute myeloid leukemia (AML): a survey of 161 cases from the French AML Intergroup. Blood. 2002 May 15;99(10):3517-23. doi: 10.1182/blood.v99.10.3517. PMID 11986202
- [Background] Yang DH, Lee JJ, Mun YC, Shin HJ, Kim YK, Cho SH, Chung IJ, Seong CM, Kim HJ. Predictable prognostic factor of CD56 expression in patients with acute myeloid leukemia with t(8:21) after high dose cytarabine or allogeneic hematopoietic stem cell transplantation. Am J Hematol. 2007 Jan;82(1):1-5. doi: 10.1002/ajh.20739. PMID 16986129
- [Background] Baer MR, Stewart CC, Lawrence D, Arthur DC, Byrd JC, Davey FR, Schiffer CA, Bloomfield CD. Expression of the neural cell adhesion molecule CD56 is associated with short remission duration and survival in acute myeloid leukemia with t(8;21)(q22;q22). Blood. 1997 Aug 15;90(4):1643-8. PMID 9269784
- [Background] Kolomietz E, Al-Maghrabi J, Brennan S, Karaskova J, Minkin S, Lipton J, Squire JA. Primary chromosomal rearrangements of leukemia are frequently accompanied by extensive submicroscopic deletions and may lead to altered prognosis. Blood. 2001 Jun 1;97(11):3581-8. doi: 10.1182/blood.v97.11.3581. PMID 11369654
- [Background] Kuss BJ, Deeley RG, Cole SP, Willman CL, Kopecky KJ, Wolman SR, Eyre HJ, Callen DF. The biological significance of the multidrug resistance gene MRP in inversion 16 leukemias. Leuk Lymphoma. 1996 Feb;20(5-6):357-64. doi: 10.3109/10428199609052416. PMID 8833390
- [Background] Bullinger L, Rucker FG, Kurz S, Du J, Scholl C, Sander S, Corbacioglu A, Lottaz C, Krauter J, Frohling S, Ganser A, Schlenk RF, Dohner K, Pollack JR, Dohner H. Gene-expression profiling identifies distinct subclasses of core binding factor acute myeloid leukemia. Blood. 2007 Aug 15;110(4):1291-300. doi: 10.1182/blood-2006-10-049783. Epub 2007 May 7. PMID 17485551
- [Background] Visani G, Bernasconi P, Boni M, Castoldi GL, Ciolli S, Clavio M, Cox MC, Cuneo A, Del Poeta G, Dini D, Falzetti D, Fanin R, Gobbi M, Isidori A, Leoni F, Liso V, Malagola M, Martinelli G, Mecucci C, Piccaluga PP, Petti MC, Rondelli R, Russo D, Sessarego M, Specchia G, Testoni N, Torelli G, Mandelli F, Tura S. The prognostic value of cytogenetics is reinforced by the kind of induction/consolidation therapy in influencing the outcome of acute myeloid leukemia--analysis of 848 patients. Leukemia. 2001 Jun;15(6):903-9. doi: 10.1038/sj.leu.2402142. PMID 11417475
- [Background] Burnett AK, Goldstone AH, Stevens RM, Hann IM, Rees JK, Gray RG, Wheatley K. Randomised comparison of addition of autologous bone-marrow transplantation to intensive chemotherapy for acute myeloid leukaemia in first remission: results of MRC AML 10 trial. UK Medical Research Council Adult and Children's Leukaemia Working Parties. Lancet. 1998 Mar 7;351(9104):700-8. doi: 10.1016/s0140-6736(97)09214-3. PMID 9504514
- [Background] Suciu S, Mandelli F, de Witte T, Zittoun R, Gallo E, Labar B, De Rosa G, Belhabri A, Giustolisi R, Delarue R, Liso V, Mirto S, Leone G, Bourhis JH, Fioritoni G, Jehn U, Amadori S, Fazi P, Hagemeijer A, Willemze R; EORTC and GIMEMA Leukemia Groups. Allogeneic compared with autologous stem cell transplantation in the treatment of patients younger than 46 years with acute myeloid leukemia (AML) in first complete remission (CR1): an intention-to-treat analysis of the EORTC/GIMEMAAML-10 trial. Blood. 2003 Aug 15;102(4):1232-40. doi: 10.1182/blood-2002-12-3714. Epub 2003 Apr 24. PMID 12714526